CLINICAL TRIAL: NCT02428439
Title: Genetic Markers and Predictors of Antidepressant-induced Suicidality in Youth Depression
Brief Title: Identification of Genetic Markers and Predictors of Antidepressant-induced Suicidality in Youth Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyo-Won Kim, Assistant professor, department of psychiatry, Asan Medical Center, Asan Medical Center
Other Study IDs: S2015-0305-0003
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Depression; Suicidal Ideation
Keywords: genetic markers; predictors; Antidepressive Agents; Suicidal Ideation; Adolescent
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Bupropion; Lamotrigine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample for GWAS(Genome-Wide Association Study)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Increased suicidality: Increase in suicidal ideation after taking the standardized pharmacotherapy (bupropion or lamotrigine) during 8 weeks.
  Interventions: Drug: bupropion or lamotrigine
- Non-increased suicidality: Non-increase of suicidal ideation after taking the standardized pharmacotherapy (bupropion or lamotrigine) during 8 weeks.
  Interventions: Drug: bupropion or lamotrigine

INTERVENTIONS:
Drug: bupropion or lamotrigine — Participants who take the standardized pharmacotherapy (bupropion or lamotrigine) for depression will be observed for 8 weeks. Drugs using in this study are the standard treatment for depression, and are NOT administered as part of this study.
  Other Names: Wellbutrin; Lamictal

SUMMARY:
The objective of this study is to identification of genetic markers and predictors of antidepressant-induced suicidality in youth depression. Participants who take the standardized pharmacotherapy (bupropion or lamotrigine) for depression will be observed for 8 weeks. They will do several scales and genetic tests at visit 1 (week 0), visit 3 (week 4) and visit 4 (week 8)

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 11 and 18 years
2. Met the Kiddie-Schedule for Affective Disorders and Schizophrenia-Present and Lifetime Version (K-SADS-PL) diagnostic criteria for depressive episode or dysthymia
3. Intelligence quotient higher than 70 on the Korean Educational Developmental Institute's Wechsler Intelligence Scale for Children

Exclusion Criteria:

1. presence of intellectual disability
2. presence of hereditary disorder
3. past and/or current history of acquired brain injury, like cerebral palsy
4. presence of seizure, other neurological disorder or sensory impairments
5. past and/or current history of pervasive developmental disorder
6. past and/or current history of schizophrenia, bipolar disorder or psychosis
7. presence of severe learning disorder

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents between 11 years and 18 years in depressed psychiatric outpatients.
  increased suicidal ideation: 14 people, non-increased suicidal ideation: 54 people, patient drop-out rate: 20%, total 80 people.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Suicidal ideation and behavior | 8 weeks
  Using Columbia-Suicide Severity Rating Scale(C-SSRS)

SECONDARY OUTCOMES:
Evaluation of treatment effect of antidepressants(CDRS) | 8 weeks
  A composite measure consisting of Children's Depression Rating scale(CDRS). Modeled after the Hamilton Rating Scale for Depression, the CDRS is a clinical interview tool designed for assessing 6-12 year-olds, and it has also been used successfully for adolescents.
Evaluation of treatment effect of antidepressants (YMRS) | 8 weeks
  A composite measure consisting of Young Mania Rating Scale(YMRS). The YMRS is an 11-item scale used to assess the severity of mania in children and adolescents ages 5-17.The YMRS has been used in clinical practice since 1978. Ratings are based on child/adolescent self-reporting and clinician observation. This instrument does not assess depressed mood.
Evaluation of treatment effect of antidepressants(P-GBI) | 8 weeks
  The P-GBI is adapted from the General Behavior Inventory, and allows parents to rate depressive, hypomanic, manic, and alternating mood symptoms in their children and adolescents ages 5-17.
Evaluation of treatment effect of antidepressants(CGI-S) | 8 weeks
  The Clinical Global Impression rating scales(CGI-S) are commonly used measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders.
Genome wide association analysis | 8 weeks
  KNIH Biobank Array

CONTACTS AND LOCATIONS:
Overall Officials: Hyowon Kim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No